CLINICAL TRIAL: NCT05074108
Title: Adapted Total Force Kitchen Pilot Intervention to Mitigate and Prevent Disordered Eating in Transitioning Service Members
Brief Title: Mitigating and Preventing Disordered Eating in Transitioning Service Members
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Not funded
Sponsor: Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Collaborators: VA Connecticut Healthcare System (U.S. Federal Agency); Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MEM-91-12005
Record Dates: First submitted 2021-08-09; First posted 2021-10-12 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2021-08

CONDITIONS: Diet, Food, and Nutrition; Healthy Eating; Eating Habit; Mindfulness
MeSH Terms: conditions — Feeding Behavior | interventions — Pilot Projects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pilot study (Experimental): Adapt and pilot a nutrition-based intervention. The program will take a holistic approach to educate participants about basic nutrition and cooking skills, sleep, and mindfulness strategies to enhance mental health.
  Interventions: Behavioral: Pilot study

INTERVENTIONS:
Behavioral: Pilot study — Aiming for an interaction 6 week course that will discuss many aspects of health and wellness.

SUMMARY:
Despite documented evidence of disordered eating (DE) among Active Duty (AD) Service Members (SM) and Veterans, DE has not been assessed in SM undergoing the transition from AD to Veterans status (AD-VS). The objective of the current study is to explore gender differences and associations between nutrition knowledge, DE attitudes and behaviors, mental health, and military-specific experiences in women and men undergoing the AD-VS transition, and then use this information along with qualitative feedback from focus groups to inform adaptations of an existing nutrition education program for pilot testing in AD-VS women and men.

DETAILED DESCRIPTION:
Despite documented evidence of disordered eating (DE) among Active Duty (AD) Service Members (SM) and Veterans, DE has not been assessed in SM undergoing the transition from AD to Veterans status (AD-VS). DE describes psychologically-driven, subclinical, maladaptive eating behaviors that do not meet diagnostic criteria for eating disorders (ED), which are serious psychiatric conditions that require intensive medical intervention and treatment. DE, while less clinically severe than ED, likely affects a much larger proportion of individuals and often goes unreported and/or underdiagnosed, thereby paving the way for chronic DE and development of deleterious outcomes. Mental health is intimately connected with eating behaviors and associations between DE/ED and other mental comorbidities have been described in AD and Veteran populations. By addressing DE during the AD-VS transition time, it may be possible to mitigate the long term clinical consequences that result from chronic DE. The AD-VS time frame is an especially opportune time to intervene with health-focused interventions given the evidence of weight gain and reductions in physical activity that occurs following separation from AD service. The contribution of DE behaviors to weight gain during and immediately following the AD-VS transition has not been explored and could be one factor to target in order to improve healthy lifestyle behaviors during this critical juncture. Interventions that provide SM with resources and strategies to prevent or minimize DE behaviors and improve mental health early in the AD-VS transition process may help to prevent adverse outcomes for Veterans. Based on the available evidence linking DE and mental health in Veterans, interventions that are able to address these issues holistically and prevent downstream clinical outcomes are worthy of investigation in AD-VS women and men. Thus, the objective of the current study is to explore gender differences and associations between nutrition knowledge, DE attitudes and behaviors, mental health, and military-specific experiences in women and men undergoing the AD-VS transition, and then use this information along with qualitative feedback from focus groups to inform adaptations of an existing nutrition education program for pilot testing in AD-VS women and men. Ultimately, this study is the first step in determining a strategy to attenuate the deleterious mental and physical health impacts of poor nutrition and DE in Veterans.

ELIGIBILITY:
Inclusion Criteria:

* Current Active Duty Service Member in the process of transitioning (e.g. separating or retiring) from the military assigned to Naval Support Activity Bethesda
* Age ≥17 years old
* Read and write English

Exclusion Criteria:

* Self-reported current or recent (past 5 years) diagnosis of a Diagnostic and Statistical Manual- (DSM-5) eating disorder including: Anorexia Nervosa, Bulimia Nervosa, or Binge Eating Disorder AND/OR
* A score of ≥15 on the Eating Disorder Examination-Questionnaire Short (EDE-QS)

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Nutrition knowledge | Pre and Post intervention, approximately 6 weeks apart
  Scores on Abridged Nutrition for Sport Knowledge Questionnaire. Questionnaire is 35 questions long. Answers are scored as either correct or incorrect. Scores range from 0-35, higher scores are more desirable and indicate greater nutrition knowledge.
Eating attitudes / behaviors | Pre and Post intervention, approximately 6 weeks apart
  Scores on Eating Pathology Symptoms Inventory. The Eating Pathology Symptoms Inventory (EPSI) is a self-report questionnaire that includes 45 items covering 8 subscales: Body Dissatisfaction, Binge Eating, Cognitive Restraint, Purging, Restricting, Excessive Exercise, Negative Attitudes toward Obesity, and Muscle Building. Each item is scored on a 5-point Likert-style scale (0 = Never; 4= Often) to describe how well each item describes the participant's experiences. Scores are derived by summing responses across the questions included in each subscale. Scores range from 0-180. Lower scores are more desirable.
Eating attitudes / behaviors | Pre and Post intervention, approximately 6 weeks apart
  Scores on Eating Disorder Examination-Questionnaire Short. The Eating Disorder Examination - Questionnaire Short (EDE-QS) was developed as a 12-item version of the Eating Disorder Examination Questionnaire (EDE-Q) with a 4-point response scale that assesses eating disorder (ED) symptoms over the preceding 7 days. Scores range from 0-36. Lower scores are more desirable.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan M Scott, PhD, Principal Investigator — Uniformed Services University of the Health Sciences

IPD SHARING:
Plan to Share IPD: No
Data generated under the funding award will be provided to the Military Women's Health Research Consortium and the Uniformed Services University, as requested in the Funding Opportunity Announcement. More broadly, data will be shared in an aggregated form through abstracts and presentations submitted to research conferences and manuscripts written for publication in peer-reviewed scientific journals. To protect the confidentiality of the participants, no data will ever be identified in publications/presentations.